CLINICAL TRIAL: NCT01876953
Title: Phase I/II Study of the Combination of Dasatinib With Chemotherapy for High Risk Acute Myeloid Leukemia (AML) Patients
Brief Title: Dasatinib, Cytarabine, and Idarubicin in Treating Patients With High-Risk Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the budget issues, the study discontinued at Phase II.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12393; NCI-2013-01141 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasatinib 100mg/day + Cytarabine 200mg/m2/day + Idarubicin 12mg/m2/day (Experimental): Patients receive cytarabine IV continuously over 168 hours on days 1-7, dasatinib PO QD on days 1-7, and idarubicin hydrochloride IV on days 1-3. Patients with non-responsive disease on day 30 may receive a second course of therapy (re-induction therapy) within 1 week in the absence of unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: dasatinib; Other: laboratory biomarker analysis
- Dasatinib 140mg/day + Cytarabine 200mg/m2/day + Idarubicin 12mg/m2/day (Experimental): Patients receive cytarabine IV continuously over 168 hours on days 1-7, dasatinib PO QD on days 1-7, and idarubicin hydrochloride IV on days 1-3. Patients with non-responsive disease on day 30 may receive a second course of therapy (re-induction therapy) within 1 week in the absence of unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: dasatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of dasatinib when given together with cytarabine and idarubicin hydrochloride and to see how well they work in treating patients with acute myeloid leukemia that is likely to come back or spread. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and idarubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving dasatinib together with cytarabine and idarubicin hydrochloride may be a better treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Of the dose levels studied, to determine the maximum tolerated dose of dasatinib when given in combination with cytarabine and idarubicin for treatment of high risk acute myeloid leukemia (AML). (Phase I)

II. To determine the anti-tumor activity of dasatinib when given in combination with cytarabine and idarubicin, as assessed by complete remission rate (CR) and remission duration. (Phase II)

SECONDARY OBJECTIVES:

I. To document CR and survival outcomes (overall, event-free). (Phase I)

II. To estimate the survival probabilities (overall and event-free) and cumulative incidence of relapse/progression. (Phase II)

III. To describe and summarize all toxicities by organ and severity. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of dasatinib, followed by a phase II study.

Patients receive cytarabine intravenously (IV) continuously over 168 hours on days 1-7, dasatinib orally (PO) once daily (QD) on days 1-7, and idarubicin hydrochloride IV on days 1-3. Patients with non-responsive disease on day 30 may receive a second course of therapy (re-induction therapy) within 1 week in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 2 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AML meeting one of the following criteria:

  * Newly diagnosed, age 60 and older
  * High risk cytogenetics and molecular abnormalities (National Comprehensive Cancer Network [NCCN] criteria)
  * Relapsed or refractory to prior chemotherapy
  * Secondary AML
* Any prior chemotherapy must have been completed >= 2 weeks prior to day 1 of study treatment and the participant must have recovered to eligibility levels from prior toxicity

  * Only one prior regimen is allowed for relapsed AML patients; note one prior regimen is defined as follows:

    * Induction chemotherapy followed by consolidation is considered one regimen
    * Induction chemotherapy followed by re-induction in case of persistent disease followed by consolidation is considered one regimen
  * Hydroxyurea is allowed prior to day 1 of study treatment to keep white blood cell (WBC) below 20 K
* Karnofsky performance status >= 60%
* Total bilirubin < 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine < 1.5 x institutional upper limit or normal OR creatinine clearance >= 60 mL/min for patients with creatinine levels above 1.5 x institutional upper limit of normal
* Ejection fraction (EF) >= 45%
* Ability to understand and sign a written informed consent document
* Patients should not be receiving any other investigational agents

Exclusion Criteria:

* Patients with clinically significant illness which would compromise participation in the study, including, but not limited to: active or uncontrolled infection, immune deficiencies or confirmed diagnosis of human immunodeficiency virus (HIV) infection, active hepatitis B, active hepatitis C, or uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmias; or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with additional (other than AML) currently active primary malignancy other than curatively treated carcinoma in situ (CIS) of the cervix, or basal or squamous cell carcinoma of the skin; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy and disease free from prior malignancies for > 2 years
* Patients with active central nervous system (CNS) disease
* Patients with Chronic Myelogenous Leukemia (CML) in Myeloid blasts crisis
* Active infections, including opportunistic infections
* Women of childbearing potential (WOCBP) who have a positive serum pregnancy test within 14 days of the first administration of oral dasatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aribi, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the funding issue, the study was stopped early before reaching the target accrual. However, all the enrolled patients had received the treatment drug per protocol.
Period: Overall Study
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
Started | 17 | 3
Completed | 17 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Total
Number analyzed (Participants) | 17 | 3 | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [27 to 73] | 63 [52 to 69] | 63 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 13 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 15 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 1 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Dasatinib (Phase I)
Description: Maximum tolerated dose of dasatinib, determined according to incidence of dose limiting toxicity (DLT), graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I)
Time Frame: From the first dose of Dasatinib through the DLT observation period (Day +28)
Population: Six patients treated at 100 mg/m2 in Phase I are evaluable for dose limiting toxicity.
Measure: Number; unit: mg/m2
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
Number analyzed (Participants) | 6
mg/m2 | 100

2. Primary Outcome: Complete Remission Rate (Phase II)
Description: Remission rates will be calculated as the percent of evaluable patients that have a confirmed CR, and exact 95% confidence intervals will be calculated for these estimates.
Time Frame: From the first cycle up to two years
Population: The study was terminated before the data were mature enough to estimate the CR rate. Therefore, the overall number of participants who were evaluable is zero.
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (Phase II)
Description: Overall survival was measured from the first dose of Dasatinib to death from any cause or last contact, whichever comes first. It was estimated using the product-limit method of Kaplan and Meier.
Time Frame: Time from start of study therapy until death, or last contact, whichever comes first, assessed up to 2 years
Population: The study was terminated before the data were mature enough to estimate the overall survival outcomes. Therefore, the overall number of participants who were evaluable is zero.
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Event-free Survival (Phase II)
Description: Event-free survival was defined as time from the first dose of Dasatinib to relapse/progression, receipt of anti-leukemia therapy, death, or last contact, whichever comes first. It was estimated using the product-limit method of Kaplan and Meier.
Time Frame: Time from start of study therapy until death, relapse/progression, receipt of anti-leukemia therapy, or last contact, whichever comes first, assessed up to two years.
Population: The study was terminated before the data were mature enough to estimate the even-free survival. Therefore, the overall number of participants who were evaluable is zero.
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event and vital status data were captured from the initial treatment to off study, up to 2 years.
Description: From day 1 to day 30, the highest grade of non-hematologic toxicities were collected. For hematologic adverse events, from day 1 to day 30, collect every grade change for hematologic toxicities grade 3 and above. After the completion of treatment, report only the worst grade of each AE and only report AEs that are possibly, probably, or definitely related to Dasatinib.
Arm/Group | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day
All-Cause Mortality (participants affected / at risk) | 11/17 | 3/3
Serious Adverse Events (participants affected / at risk) | 4/17 | 0/3
Other Adverse Events (participants affected / at risk) | 17/17 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day (N=17) | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day (N=3)
Death NOS (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day (N=17) | Dasatinib 140mg/Day + Cytarabine 200mg/m2/Day + Idarubicin 12mg/m2/Day (N=3)
10002272-Anemia (Blood and lymphatic system disorders) | 16 (83) | 3 (3)
10016288-Febrile neutropenia (Blood and lymphatic system disorders) | 5 (12) | 0 (0)
Markedly irregular multilobulated spleen with linear calcification (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
10003658-Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
10003662-Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
10034474-Pericardial effusion (Cardiac disorders) | 1 (2) | 2 (2)
10040741-Sinus bradycardia (Cardiac disorders) | 6 (12) | 0 (0)
10040752-Sinus tachycardia (Cardiac disorders) | 12 (34) | 1 (1)
Atherosclerotic Vascular Disease (Cardiac disorders) | 0 (0) | 1 (1)
Left atrial enlargment (Cardiac disorders) | 0 (0) | 1 (1)
Nonspecific ST and T wave abnormality (Cardiac disorders) | 1 (1) | 0 (0)
cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
10065837-External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Mastoiditis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
right ear hearing loss (Ear and labyrinth disorders) | 1 (3) | 0 (0)
syndrome of inappropriate antidiuretic hormone (Endocrine disorders) | 1 (1) | 0 (0)
10005886-Blurred vision (Eye disorders) | 1 (1) | 0 (0)
10013774-Dry eye (Eye disorders) | 2 (4) | 1 (1)
10047848-Watering eyes (Eye disorders) | 1 (1) | 0 (0)
redness, jaundice, sclera/conjunctiva discoloration (Eye disorders) | 0 (0) | 1 (1)
scleral hemmorage (Eye disorders) | 1 (1) | 0 (0)
scleral hemorage (Eye disorders) | 1 (1) | 0 (0)
10000060-Abdominal distension (Gastrointestinal disorders) | 3 (4) | 0 (0)
10000081-Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
10003445-Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
10009887-Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
10010774-Constipation (Gastrointestinal disorders) | 7 (10) | 1 (1)
10012727-Diarrhea (Gastrointestinal disorders) | 12 (24) | 3 (3)
10013781-Dry mouth (Gastrointestinal disorders) | 5 (8) | 0 (0)
10013946-Dyspepsia (Gastrointestinal disorders) | 3 (5) | 1 (1)
10013950-Dysphagia (Gastrointestinal disorders) | 4 (5) | 0 (0)
10015388-Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
10016296-Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
10017999-Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
10018286-Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
10019611-Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
10028130-Mucositis oral (Gastrointestinal disorders) | 9 (21) | 2 (2)
10028813-Nausea (Gastrointestinal disorders) | 13 (27) | 3 (3)
10031009-Oral pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
10038072-Rectal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
10044055-Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
10047700-Vomiting (Gastrointestinal disorders) | 9 (12) | 0 (0)
10055356-Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernias (Gastrointestinal disorders) | 0 (0) | 1 (1)
10008531-Chills (General disorders) | 4 (5) | 0 (0)
10014222-Edema face (General disorders) | 2 (3) | 0 (0)
10016059-Facial pain (General disorders) | 1 (1) | 0 (0)
10016256-Fatigue (General disorders) | 10 (26) | 3 (3)
10016558-Fever (General disorders) | 13 (36) | 2 (3)
10017577-Gait disturbance (General disorders) | 1 (1) | 0 (0)
10022095-Injection site reaction (General disorders) | 1 (1) | 0 (0)
10025482-Malaise (General disorders) | 1 (1) | 1 (1)
10033371-Pain (General disorders) | 4 (5) | 0 (0)
10050068-Edema limbs (General disorders) | 9 (17) | 3 (3)
10051792-Infusion related reaction (General disorders) | 1 (1) | 0 (0)
10062466-Localized edema (General disorders) | 1 (1) | 0 (0)
10062501-Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
generalized edema (General disorders) | 1 (2) | 0 (0)
biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
10007810-Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
10019799-Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
10040047-Sepsis (Infections and infestations) | 2 (2) | 0 (0)
10040753-Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
10048038-Wound infection (Infections and infestations) | 1 (2) | 0 (0)
10048762-Tooth infection (Infections and infestations) | 1 (2) | 0 (0)
10061229-Lung infection (Infections and infestations) | 2 (3) | 1 (1)
10062255-Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
10069138-Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Candida Glabrata (Infections and infestations) | 0 (0) | 1 (1)
Enterococci Faecium (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis Grade 1 CT scan dated 10/9 (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus Coagulase Negative (Infections and infestations) | 0 (0) | 1 (1)
Streptococcus viridans bacteremi (Infections and infestations) | 1 (1) | 0 (0)
Upper lip herpetic lesion (Infections and infestations) | 0 (0) | 1 (1)
10006504-Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
10016173-Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
10000636-Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
10001551-Alanine aminotransferase increased (Investigations) | 9 (12) | 2 (2)
10001675-Alkaline phosphatase increased (Investigations) | 6 (7) | 2 (2)
10003481-Aspartate aminotransferase increased (Investigations) | 9 (16) | 1 (1)
10005364-Blood bilirubin increased (Investigations) | 11 (34) | 3 (3)
10007612-Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
10011368-Creatinine increased (Investigations) | 5 (5) | 0 (0)
10022402-INR increased (Investigations) | 0 (0) | 1 (1)
10025256-Lymphocyte count decreased (Investigations) | 15 (44) | 3 (3)
10025258-Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
10029366-Neutrophil count decreased (Investigations) | 12 (24) | 3 (3)
10035528-Platelet count decreased (Investigations) | 17 (119) | 3 (3)
10047896-Weight gain (Investigations) | 6 (13) | 2 (2)
10047900-Weight loss (Investigations) | 9 (17) | 1 (1)
10049182-White blood cell decreased (Investigations) | 16 (37) | 1 (1)
10050528-Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
10056910-GGT increased (Investigations) | 1 (1) | 0 (0)
10000486-Acidosis (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
10001680-Alkalosis (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
10002646-Anorexia (Metabolism and nutrition disorders) | 10 (19) | 2 (2)
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
10020680-Hypernatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
10020907-Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (49) | 3 (3)
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 12 (25) | 2 (2)
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
10021018-Hypokalemia (Metabolism and nutrition disorders) | 12 (42) | 3 (3)
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
10021038-Hyponatremia (Metabolism and nutrition disorders) | 16 (37) | 2 (2)
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 6 (9) | 0 (0)
10029883-Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10003246-Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 7 (13) | 3 (4)
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5)
10048706-Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
10012373-Depressed level of consciousness (Nervous system disorders) | 1 (3) | 0 (0)
10013911-Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
10019211-Headache (Nervous system disorders) | 9 (22) | 1 (1)
10024264-Lethargy (Nervous system disorders) | 2 (2) | 0 (0)
10027175-Memory impairment (Nervous system disorders) | 3 (3) | 0 (0)
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
10039906-Seizure (Nervous system disorders) | 2 (2) | 0 (0)
10041349-Somnolence (Nervous system disorders) | 3 (4) | 0 (0)
10044565-Tremor (Nervous system disorders) | 1 (1) | 0 (0)
seizure-like disorder, altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
10001497-Agitation (Psychiatric disorders) | 4 (6) | 1 (1)
10002855-Anxiety (Psychiatric disorders) | 7 (12) | 0 (0)
10010300-Confusion (Psychiatric disorders) | 3 (3) | 1 (1)
10012378-Depression (Psychiatric disorders) | 2 (2) | 1 (1)
10022437-Insomnia (Psychiatric disorders) | 5 (14) | 3 (3)
10038743-Restlessness (Psychiatric disorders) | 4 (7) | 0 (0)
10019450-Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
10037032-Proteinuria (Renal and urinary disorders) | 3 (3) | 1 (1)
10046539-Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
10046543-Urinary incontinence (Renal and urinary disorders) | 3 (3) | 0 (0)
10069339-Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
10013934-Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
10018146-Genital edema (Reproductive system and breast disorders) | 2 (7) | 0 (0)
10039757-Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
10046912-Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Thickened Endometrium (Reproductive system and breast disorders) | 1 (1) | 0 (0)
10003598-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 1 (1)
10020201-Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
10021143-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
10035598-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
10035623-Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
10035742-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
10036402-Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10036790-Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
10037375-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10037400-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10040975-Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
10047924-Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Bilateral lower lobe interstitial changes possible infiltrates. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LLL infiltrate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peribronchial infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right bundle branch block (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chest infiltrate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
vascular congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
10037847-Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (25) | 3 (3)
10040865-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
10040947-Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
10051837-Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
10054524-Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
10054541-Periorbital edema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
blisters (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
desquamation in both hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nasal lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
petechial rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
10007196-Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
10016825-Flushing (Vascular disorders) | 3 (3) | 0 (0)
10019428-Hematoma (Vascular disorders) | 1 (1) | 0 (0)
10020772-Hypertension (Vascular disorders) | 16 (100) | 3 (4)
10021097-Hypotension (Vascular disorders) | 4 (10) | 0 (0)
10043565-Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT01876953/Prot_SAP_000.pdf